CLINICAL TRIAL: NCT03231592
Title: Im(Proving) the CSA Model
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Community Health Center of Franklin County (Other)
Collaborators: Just Roots (Unknown); Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FMPP2016
Record Dates: First submitted 2017-05-09; First posted 2017-07-27 (Actual); Last update posted 2017-07-27 (Actual); Status verified 2017-07

CONDITIONS: Overweight and Obesity; Nutrition Poor; Diet Modification
MeSH Terms: conditions — Overweight; Obesity; Malnutrition

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CSA Group (Experimental): This group will receive CSA Shares (a selection of fresh fruits and vegetables from a local farm) each week for 24 weeks over the summer of 2017 and 2018. The CSA does not operate over the winter.
  Interventions: Other: CSA Group
- Enhanced Usual Care Group (Active Comparator): This group will receive a handout about healthy eating, in addition to routine care in their primary care practice.
  Interventions: Other: Enhanced Usual Care Group

INTERVENTIONS:
Other: CSA Group — Already included in the arm descriptions.
  Arms: CSA Group
Other: Enhanced Usual Care Group — Already included in the arm descriptions.
  Arms: Enhanced Usual Care Group

SUMMARY:
In 1986, The Pioneer Valley in Western Massachusetts was home to one of the first two community supported agriculture (CSA) businesses in the USA. In 2014, there were 6,200 CSAs across the states, and today, in the Pioneer Valley alone, there are sixty CSAs. As with many parts of the United States, there are too many CSAs competing for the same pool of middle and upper-class customers. In his research at the University of Massachusetts in 2014, Mark Paul stated CSA farms are trapped in a lose-lose conundrum in which the farmers are not making enough money for a living wage, while simultaneously CSA shares are too expensive for many community members. The central challenge facing the CSA model moving forward is to provide fair compensation to farmers and farm workers, while making shares available at prices that can attract more members of the community. "(Im)Proving the CSA Model" proposes to increase consumption of and access to local products AND to develop new market opportunities for farms by opening the CSA membership base nationwide to low-income consumers and more price conscious middle class consumers. The investigators will do this by researching and documenting the health benefits of belonging to a CSA program. The investigators expect the resulting data to justify insurance-provided cash "wellness" benefits for CSA participation, much like those currently provided for gym membership. A wellness benefit will provide the financial incentive necessary to open CSA programs to lower- and middle-income consumers.

The two-year research study intends to demonstrate that enrolling community health center patients in a Community Supported Agriculture (CSA) program is feasible and leads to dietary improvements that would be expected to offer clinical benefits in larger scale studies over longer timeframes. To maximize the knowledge gained from participation in this study, the investigators will measure several self-reported, laboratory, and clinical outcomes, but the primary purpose of this study is to provide pilot data for the model.

To test this the investigators will implement a randomized controlled clinical trial design, with individual-level randomization of 120 participants, assigned in 1:1 ratio to receipt of a CSA membership (goal: 60 participants) or enhanced usual care (goal: 60 participants).

DETAILED DESCRIPTION:
Full study protocol is available upon request from Rochelle Bellin

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* BMI > 25 kg/m2 in the past 1 year
* Willing to commit to random assignment to either receive CSA membership or enhanced care control
* Stable health, with no severe medical comorbidities that might interfere with their ability to participate in the intervention, such as severe psychiatric illness or imminent hospitalization
* Be willing to keep a food diary for one week
* Be willing to attend and complete 5 examinations
* Be able to understand and communicate effectively in English
* Ability to store and prepare food

Exclusion Criteria:

* Must not be pregnant or planning pregnancy in the next year
* Currently enrolled in another study of dietary quality
* Life threatening food allergy to component of CSA boxes
* Currently enrolled in other CSA, or planning to enroll in CSA if assigned to enhanced usual care control group

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2017-05-10 (Actual); Primary Completion 2018-12-20 (Estimated); Study Completion 2018-12-20 (Estimated)

PRIMARY OUTCOMES:
HEI2010 Score | 19 months
  The HEI 2010 score is an indicator of dietary quality.

SECONDARY OUTCOMES:
Health Related Quality of Life | 19 months
  We will use the PROMIS-10 Global Health instrument to assess Health Related Quality of Life

OTHER OUTCOMES:
Estimate the return on investment of CSA membership | 19 months
  To estimate the return on investment of CSA membership. We will use effects on dietary quality and quality of life obtained from Outcome 1 and employ an existing microsimulation model of health expenditures to determine the change in health expenditures attributable to program participation divided by the costs of the program to calculate the 'return on investment'. The focus of our analysis will be identifying health effects that are relevant to accountable care organizations and insurers with the goal of informing adoption of the CSA model.
BMI | 19 months
  Body Mass Index. This is an exploratory outcome and the study is not necessarily powered to detect changes
Blood Pressure | 19 months
  Systolic and Diastolic Blood Pressure. This is an exploratory outcome and the study is not necessarily powered to detect changes
Hemoglobin A1c | 19 months
  Hemoglobin A1c. This is an exploratory outcome and the study is not necessarily powered to detect changes
Lipids | 19 months
  Non-fasting lipid panels (including total cholesterol, HDL, triglycerides, and LDL if calculable). This is an exploratory outcome and the study is not necessarily powered to detect changes
Food Insecurity | 19 months
  USDA Food Security Survey module, 10 adult referenced items, modified to have a 1 month look back period, using standard scoring. This is an exploratory outcome and the study is not necessarily powered to detect changes
Anxiety Symptoms | 19 months
  Measured using the PROMIS Emotional Distress Anxiety 4 item short-form.This is an exploratory outcome and the study is not necessarily powered to detect changes
Depressive Symptoms | 19 months
  Measured using the PROMIS Emotional Distress Depression 4 item short-form. This is an exploratory outcome and the study is not necessarily powered to detect changes
Cost Related Medication Underuse | 19 months
  Measured using the 4 cost-related medication underuse items from MEPS/NHISThis is an exploratory outcome and the study is not necessarily powered to detect changes
Food-Medication Trade-Offs | 19 months
  4 questions about trade-offs between affording food, medications, and meeting other basic needs. This is an exploratory outcome and the study is not necessarily powered to detect changes

CONTACTS AND LOCATIONS:
Overall Officials: Edward Sayer, Principal Investigator — Community Health Center of Franklin County
Locations (1):
- Community Health Center of Franklin County, Greenfield, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Berkowitz SA, O'Neill J, Sayer E, Shahid NN, Petrie M, Schouboe S, Saraceno M, Bellin R. Health Center-Based Community-Supported Agriculture: An RCT. Am J Prev Med. 2019 Dec;57(6 Suppl 1):S55-S64. doi: 10.1016/j.amepre.2019.07.015. Epub 2019 Sep 12. PMID 31522922
- See also: 24-hour dietary recall tool to be used at each Research Visit to assess participants previous 24 hours of consumption — https://asa24.nci.nih.gov/